CLINICAL TRIAL: NCT01600443
Title: A Randomized Cross-over Study on Urethral Microtrauma After Intermittent Catheterization.
Brief Title: Comparison of Microtrauma in Urethra After Usage of Different Catheters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned interim analysis showed study was underpowered
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOF-0022
Record Dates: First submitted 2012-04-24; First posted 2012-05-17 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Hematuria
MeSH Terms: conditions — Hematuria

ARMS (6):
- LoFric - SC - SCCM (Experimental): Study period 1: LoFric Study period 2: SpeediCath Study period 3: SpeediCath Compact Male In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male
- LoFric - SCCM - SC (Experimental): Study period 1: LoFric Study period 2: SpeediCath Compact Male Study period 3: SpeediCath In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male
- SC - SCCM - LoFric (Experimental): Study period 1: SpeediCath Study period 2: SpeediCath Compact Male Study period 3: LoFric In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male
- SC - LoFric - SCCM (Experimental): Study period 1: SpeediCath Study period 2: LoFric Study period 3: SpeediCath Compact Male In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male
- SCCM - LoFric - SC (Experimental): Study period 1: SpeediCath Compact Male Study period 2: LoFric Study period 3: SpeediCath In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male
- SCCM - SC - LoFric (Experimental): Study period 1: SpeediCath Compact Male Study period 2: SpeediCath Study period 3: LoFric In each study period three catheterizations are made, separated by at least 2 hours.
  Interventions: Device: LoFric; Device: SpeediCath; Device: SpeediCath Compact Male

INTERVENTIONS:
Device: LoFric — Three catheterizations at least two hours apart using LoFric Primo 40 cm CH14.
Device: SpeediCath — Three catheterizations at least two hours apart using SpeediCath 40 cm CH14.
Device: SpeediCath Compact Male — Three catheterizations at least two hours apart using SpeediCath Compact Male 30 cm.

SUMMARY:
The study is undertaken to investigate if the urethral microtrauma, caused by intermittent catheterization, differs between three hydrophilic catheters for intermittent catheterization, LoFric; SpeediCath (SC) and SpeediCath Compact Male (SCCM). The study is a prospective, randomised, cross-over, single-centre study.

Each subject will be randomized to use three different catheter types. Three catheterizations will be performed with each catheter type during one day, with at least two hours between each catheterization. The washout period between catheter switch will be at least one week.

The primary objective is to evaluate urethral microtrauma for three hydrophilic catheters with regards to hematuria after intermittent catheterization.

The secondary objectives are to evaluate urethral microtrauma for three hydrophilic catheters with regards to pyuria and subjective evaluation after intermittent catheterization.

The safety of the three catheters will be evaluated in terms of adverse advents, non-serious and serious, rated for causality.

The hypothesis that level of hematuria is equal after using different catheters will be tested using Wilcoxon signed rank test. The hypothesis will be rejected if the p-value is less than 5%.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Healthy male volunteers aged 18 years and over (half of the included subjects shall be 18-50 years and the other half >50 years old)
3. Negative urine dipstick test (no blood in the urine) before randomization

Exclusion Criteria:

1. Intake of anticoagulants at enrolment and during the study period
2. Intake of antibiotics at enrolment and during the study period
3. Urinary tract infection (UTI) at enrolment and during the study period
4. Known abnormalities or diseases of the lower urinary tract with the exception of BPH
5. Kidney stones
6. Tumour in the urinary tract
7. Known Sexually transferable diseases in the urinary tract during the study period
8. Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
9. Previous enrolment or randomisation of treatment in the present study
10. Simultaneous participation in another clinical study that might interfere with the endpoints of the study, as deemed by the investigator
11. Severe non-compliance to protocol as judged by the investigator and/or Astra Tech

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Hematuria | Approximately 2 hours after last catheterization
  Blood in urine (measured by microscopic urine sediment evaluation) will be assessed at the first normal micturition after three catheterizations. Comparison will be made between study catheter/visit days.

SECONDARY OUTCOMES:
Hematuria | At first, second and third catheterization, approximately 2 hours apart
  Blood in urine (measured by microscopic urine sediment evaluation). Comparison will be made between study catheter/visit days.
Pyuria | At first, second and third catheterization, approximately 2 hours apart
  White blood cells in urine (measured by microscopic urine sediment evaluation). Comparison will be made between study catheter/visit days.
Pyuria | Approximately 2 hours after last catheterization
  White blood cells in urine (measured by microscopic urine sediment evaluation) will be assessed at first normal micturition after three catheterizations. Comparison will be made between study catheter/visit days.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmkvist, Assoc Prof, Principal Investigator — Skane University Hospital
Locations (1):
- Clinical Trial Unit, R&D Centre Skåne, Skåne University Hospital, Lund, Sweden